CLINICAL TRIAL: NCT05905848
Title: Pre-operative Antihypertensive Drugs and Persistent Hypotension in Carotid Artery Stenting Comorbid With Hypertension Patients --- a Multicenter, Randomized, Open Label, Blinded Ended Point Clinic Trail
Brief Title: Pre-operative Antihypertension Strategies-Carotid Artery Stenting
Acronym: PASS-CAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Bo Wu, Professor/Deputy Director of Neurology of West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023(728)
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Carotid Stenosis
Keywords: Carotid Artery Stenting; Sinus Reflex; Antihypertensive drugs; Catecholamine
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Intervention Model Description: RASI group and CCB group
Who Masked: Outcomes Assessor
Masking Description: open label, blinded endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RASI group (Experimental): Administer RASI, with or without other antihypertensives except for CCB, and blood pressure should be controlled within the target range (140/90 mmHg). RASI intaking starts at least 5 days before stenting.
  Interventions: Drug: administering RASI (the trade name or universal name will not be stipulated) before stenting
- CCB group (Active Comparator): Administer CCB, with or without other antihypertensives except for RASI, and blood pressure should be controlled within the target range (140/90 mmHg). CCB intaking starts at least 5 days before stenting.
  Interventions: Drug: administering CCB (the trade name or universal name will not be stipulated) before stenting

INTERVENTIONS:
Drug: administering RASI (the trade name or universal name will not be stipulated) before stenting — Pre-operative antihypertensive drugs before stenting will be random assigned (RASI or CCB) at least 5 days before stenting. Patients in RASI group will receive RASI (all kinds of RASI will be permited and the trade name or universal name of drugs will not be limited), with or without other antihypertensives except for CCB (any kind of CCB).
  Blood pressure of patients should be controlled within the target range (140/90 mmHg); and usage and dosage of antihypertensive drugs will not be stipulated. Grapefruit intaking should be avoid.
  Arms: RASI group
Drug: administering CCB (the trade name or universal name will not be stipulated) before stenting — Pre-operative antihypertensive drugs before stenting will be random assigned (RASI or CCB) at least 5 days before stenting. Patients in CCB group will receive CCB (all kinds of CCB will be permited and the trade name or universal name of drugs will not be limited), with or without other antihypertensives except for RASI (any kind of RASI).
  Blood pressure of patients should be controlled within the target range (140/90 mmHg); and usage and dosage of antihypertensive drugs will not be stipulated. Grapefruit intaking should be avoid.
  Arms: CCB group

SUMMARY:
Carotid artery stenting (CAS) is one of major treatments in prevention of ischemic stroke. Because of sinus reflex due to stenting and balloon dilatation, persistent post-surgery hypotension is a common perioperative event. Persistent hypotension can lead to perioperative adverse events like ischemic stroke, myocardial infraction, renal failure and death; or more usually, it prolongs length of stay and hospital expenses. Renin-angiotensin-aldosterone inhibitor (RASI) could inhibit the release of catecholamine and may lead to higher rate of persistent hypotension after CAS compared to other hypertensives.Thus, the investigators aim to investigate the effect of pre-operation antihypertensive drugs on persistent hypotension after stenting, and followed burden in carotid artery stenting comorbid with hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* have a history of TIA or nondisabling ischemic stroke within the past 6 months (symptomatic) with ipsilateral initial part of EICA stenosis ≥ 50 % or asymptomatic with initial part of EICA stenosis ≥ 70%, and the cause of stenosis was atherosclerosis
* have hypertension requiring hypertensives
* modified Rankin scale (mRS) before stenting < 3

Exclusion Criteria:

* with ipsilateral tandem stenosis
* with history of operation in contralateral carotid artery, like stenting, endarterectomy and bypass.
* requiring operation in contralateral carotid artery in the same admission.
* requiring general anesthesia in the same operation (stenting)
* with contraindication to carotid stenting, such as Inability to tolerate surgery due to organ dysfunction, cerebral aneurism, cerebral hemorrhage in 3 months, myocardial infraction or large-area cerebral infraction within 2 weeks, extreme tortuosity of the vessel
* allergic to Calcium channel blockers, angiotensin receptor blockers or hydrochlorothiazide
* pregnancy
* with concomitant medication as following: Azole antifungals, macrolides antibiotics, cardiac calcium channel blockers, Rifampicin, sildenafil, simvastatin, immunosuppressants, antidepressants, valproic acid, cimetidine, aliskiren, NSAIDs, protease inhibitors (ritonavir) and drugs that affect potassium in the blood
* with hepatic insufficiency, renal insufficiency, kidney transplantation, diabetic nephropathy, biliary obstructive disease, or the presence of end-stage disease affecting clinical prognosis assessment (such as end-stage cancer, end-stage heart disease, liver failure, renal failure, pulmonary failure)
* with depression, schizophrenia, bipolar disorder, epilepsy, tuberculosis, AIDS, primary hyperaldosteronism, hyperkalemia, hypercalcemia, hyperuricemia, gout
* participating other trails which would affect the evaluation of outcomes
* with reserpine and clonidine intake within 1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of persistent post-surgery hypotension | the first 24 hours after CAS
  systolic blood pressure (SBP) < 90 mmHg or requiring vasopressor with lasting > 6 hours, and without evidence hypovolemia and heart failure

SECONDARY OUTCOMES:
Length of stay after surgery | From surgery to dicharge, up to 3 month.
Hospital expenses after surgery, based on payment list in hospital information system | From surgery to dicharge, up to 3 month.
  Payment list in hospital information system for all patients will be recorded with permission and the hospital expenses after surgery will be caculated based on those records.
Difference of serum catecholamine (adrenalin, norepinephrine and dopamine) before and after surgery (all in unit of nmol/L) | at morning (7 o'clock am) of the day of surgery and the first day after surgery
Difference of heart rate variability (HRV) before and after surgery | 24 hours before surgery to at least 24 hours after surgery
The incidence of bradycardia after surgery | the first 24 hours after CAS
The total incidence of stroke, myocardial infraction, renal failure and embolism of retinal arteries | From surgery to dicharge, up to 3 month.

OTHER OUTCOMES:
The total incidence of cardiac and cerebral events (stroke, myocardial infarction, heart failure and angina pectoris) and symptomatic hypotension | From administering antihypertensive drugs to stenting, at least 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wu, Dr, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Outcomes and grouping of patticipants will be shared to all investigators contributing to this study. Study protocol, statistical analysis plan will also be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 6 month after the recruitment completed